CLINICAL TRIAL: NCT06800573
Title: The Effect of Integrating a Smartphone Application with Global Postural Re-education on Cervical Proprioception in Patients with Upper Cross Syndrome
Brief Title: Smartphone Application with Global Postural Re-education in Patients with Upper Cross Syndrome
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Rania Ahmed, principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P.T.REC/012/005034
Record Dates: First submitted 2025-01-22; First posted 2025-01-30 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2025-01

CONDITIONS: Upper Cross Syndrome
MeSH Terms: conditions — Oculocerebral hypopigmentation syndrome type Preus

STUDY DESIGN:
Intervention Model Description: The Effect of Integrating a Smartphone Application with Global Postural Re-education on Cervical Proprioception in Patients with Upper Cross Syndrome
  Design:
  Randomized Controlled Trial.
  Participants:
  The sample size will be determined using G power analysis.
  Procedures:
  Patients of both sexes (men and women) suffering from cervical pain caused by Upper Cross Syndrome (UCS) will be randomly selected from El Amal Clinic in Fayoum. They will be randomly assigned into three groups:
  Group A: Participants will undergo experimental interventions for approximately 50 minutes a day, 4 days a week, for an 8-week period. Exercises will be assisted and reminded by a smartphone app at predetermined times.
  Group B: Participants will undergo the same experimental interventions for approximately 50 minutes a day, 4 days a week, for an 8-week period, without app assistance. The exercises include:
  Exercise 1: The lying posture with leg extension progression, aimed to stretch the anterior muscle c
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group A: underwent the experimental interventions about 50 min a day, 4 days a week for an 8-week (Experimental)
  Interventions: Other: smartphone app exercises
- • Group B: underwent the experimental interventions about 50 min a day, 4 days a week for an 8-week (Experimental): • Group B: underwent the experimental interventions about 50 min a day, 4 days a week for an 8-week period.
  Interventions: Other: lying posture with progression
- • control group: The participants in the performed an evidence-based physiotherapy program about 50 (Active Comparator): • control group: The participants in the performed an evidence-based physiotherapy program about 50 min a day, 4 days a week for an 8-week period, described as a postural correction on daily activities .
  Interventions: Other: Conventional physical therapy

INTERVENTIONS:
Other: Conventional physical therapy — including strengthening exercises for deep neck flexors, rhomboids, lower trapezius and serratus anterior, (2 sets of 10 repetitions per day) and stretching exercises for pectoralis muscles (20seconds hold, 5 repetition.
  Arms: • control group: The participants in the performed an evidence-based physiotherapy program about 50
Other: lying posture with progression — Exercise 1, the lying posture with leg extension progression, was aimed to stretch the anterior muscle chain (diaphragm, pectoralis minor, scalene, sternocleidomastoid, intercostalis, iliopsoas, arm, forearm, and hand flexors)(Bonetti et al., 2010).
  Exercise 2, the lying posture with flexion of the thighs, was intended to stretch the posterior chain (upper trapezius, levator scapulae, suboccipital, erector spinae, gluteus maximus, ischiotibial, triceps surae, and foot intrinsic muscles).
  Arms: • Group B: underwent the experimental interventions about 50 min a day, 4 days a week for an 8-week
Other: smartphone app exercises — about 50 min a day, 4 days a week for an 8-week period also, performed exercises which were reminded by a smartphone app at predetermined times.
  Arms: Group A: underwent the experimental interventions about 50 min a day, 4 days a week for an 8-week

SUMMARY:
The Effect of Integrating a Smartphone Application with Global Postural Re-education on Cervical Proprioception in Patients with Upper Cross Syndrome

Design:

Randomized Controlled Trial (RCT).

Procedures:

Patients with cervical pain resulting from Upper Cross Syndrome (UCS), recruited from El Amal Clinic in Fayoum, will be randomly assigned to one of three groups:

Group A: Receives experimental interventions for 50 minutes per day, 4 days per week, over 8 weeks. The exercises are assisted by a smartphone application designed to support the intervention.

Group B: Receives the same interventions as Group A but without the use of the smartphone application. The exercises focus on stretching the anterior and posterior muscle chains.

Control Group: Receives conventional physiotherapy for 50 minutes per day, 4 days per week, over 8 weeks. This includes postural correction, neck education, and exercise therapy.

Inclusion Criteria:

Office workers aged between 28 and 48 years.

Chronic nonspecific neck pain with a Visual Analog Scale (VAS) score between 3 and 8.

Persistent pain for more than 3 months.

Absence of cognitive impairments and the ability to safely participate in an exercise program.

Postural changes characteristic of UCS, such as forward head posture and elevated shoulders.

Exclusion Criteria:

Specific causes of neck pain, such as systemic diseases or neurological signs.

History of spinal surgery or physical therapy treatments within the last 6 months.

Failure to attend three consecutive sessions or four non-consecutive sessions.

Instrumentation:

Assessment Tools:

Visual Analog Scale (VAS) to measure cervical pain.

Cervical Range of Motion (CROM) device to assess cervical range of motion and proprioception.

Neck Disability Index (NDI) to evaluate neck function.

Treatment Tools:

Smartphone application named "Kyphosis and Rounded Back."

Global Postural Reeducation methods.

Traditional physiotherapy techniques.

DETAILED DESCRIPTION:
The Effect of Integrating a Smartphone Application with Global Postural Re-education on Cervical Proprioception in Patients with Upper Cross Syndrome

Design:

Randomized Controlled Trial.

Participants:

The sample size will be determined using G power analysis.

Procedures:

Patients of both sexes (men and women) suffering from cervical pain caused by Upper Cross Syndrome (UCS) will be randomly selected from El Amal Clinic in Fayoum. They will be randomly assigned into three groups:

Group A: Participants will undergo experimental interventions for approximately 50 minutes a day, 4 days a week, for an 8-week period. Exercises will be assisted and reminded by a smartphone app at predetermined times.

Group B: Participants will undergo the same experimental interventions for approximately 50 minutes a day, 4 days a week, for an 8-week period, without app assistance. The exercises include:

Exercise 1: The lying posture with leg extension progression, aimed to stretch the anterior muscle chain (diaphragm, pectoralis minor, scalene, sternocleidomastoid, intercostalis, iliopsoas, arm, forearm, and hand flexors).

Exercise 2: The lying posture with flexion of the thighs, intended to stretch the posterior chain (upper trapezius, levator scapulae, suboccipital, erector spinae, gluteus maximus, ischiotibial, triceps surae, and foot intrinsic muscles).

Control Group: Participants will perform an evidence-based physiotherapy program for approximately 50 minutes a day, 4 days a week, for an 8-week period. This program includes:

Postural correction in daily activities, neck education, and exercise therapy focused on issues such as spine anatomy, physiology, biomechanics, common causes of neck pain, the load tolerance model, nociceptive pain processing, self-care, and ergonomic suggestions for daily activities (e.g., standing, sitting, lifting).

Conventional physical therapy, including strengthening exercises for deep neck flexors, rhomboids, lower trapezius, and serratus anterior (2 sets of 10 repetitions per day) and stretching exercises for pectoralis muscles (20-second hold, 5 repetitions).

Inclusion Criteria:

Office workers using a computer for at least 4 hours per day.

Aged between 28 and 48 years.

Neck pain scored between 3 and 8 cm on a Visual Analog Scale (VAS) (0 indicating no pain and 10 indicating unbearable pain).

Chronic nonspecific neck pain lasting more than 3 months.

Willingness and ability to safely participate in an exercise program without cognitive impairments.

Specific postural changes seen in UCS, including forward head posture, increased cervical lordosis and thoracic kyphosis, elevated and protracted shoulders, and scapular rotation, abduction, or winging.

Exclusion Criteria:

Specific causes of neck pain (e.g., systemic, rheumatic, or neuromuscular diseases), central or peripheral neurological signs, cognitive impairments, spinal surgery, or physiotherapy treatments in the 6 months prior to baseline assessment.

Participants missing at least three consecutive or four non-consecutive sessions.

Instrumentation:

For Assessment:

Visual Analog Scale (VAS) to assess cervical pain.

CROM device to assess cervical range of motion (ROM) and cervical proprioception.

Neck Disability Index (NDI) to assess neck function.

For Treatment:

Smartphone app called "Kyphosis and Rounded Back" .

Global Postural Re-education.

Traditional evidence-based physiotherapy.

ELIGIBILITY:
Inclusion Criteria:

office workers(using a computer at least 4 h),

* aged between 28 and 48years,
* NP between 3 and 8 cm on a visual analog scale(VAS) (from 0 indicating no pain at all to 10 indicating unbearable pain),
* Chronic non specific neck pain lasting for more than 3 months (Fathollahnejad et al., 2019).

Exclusion Criteria:

* • Specific causes of NP (e.g., systemic, rheumatic, neuromuscular diseases), central or peripheral neurological signs, cognitive impairment, spinal surgery, or physical therapy treatments in the last 6 months prior to the baseline assessment.

  * Participants would be also excluded if they missed at least three consecutive or four non consecutive sessions (Fathollahnejad et al., 2019).

Ages: 28 Years to 48 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-03-25 (Estimated); Primary Completion 2025-07-20 (Estimated); Study Completion 2025-08-28 (Estimated)

PRIMARY OUTCOMES:
VAS (visual analogue scale) | 8 weeks
  1. VAS (visual analogue scale) to assess cervical pain.

SECONDARY OUTCOMES:
Cervical ROM | 8 weeks
  CROM device to assess cervical ROM and to assess cervical propioception.
Neck disability index (NDI) | 8 weeks
  Neck disability index (NDI): to assess neck function.